CLINICAL TRIAL: NCT06507748
Title: A Study to Evaluate the Feasibility of a Physiologic Biomarker to Assess Pain and Other Sensory Problems Using Pupillometry in Participants With Neurofibromatosis Type 1 (NF1)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 10001826; 001826-C
Record Dates: First submitted 2024-07-17; First posted 2024-07-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-22

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis Type 1; Plexiform Neurofibromas; Pain; Sensation; Clinical outcomes; Objective measurement; Biomarker
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1/Feasibility and longitudinal assessments (Other): Evaluation with the AlgometRx device and patient- and observer-reported outcome measures
  Interventions: Device: AlgometRx Nociometer

INTERVENTIONS:
Device: AlgometRx Nociometer — Novel objective pain measurement device

SUMMARY:
Background:

Neurofibromatosis type 1 (NF1) is a genetic condition that causes tumors to grow along the nerves in the skin, brain, and other parts of the body. People with NF1 often have pain and may experience other abnormal sensations like itching, numbness, or tingling. These symptoms can affect their daily life. Researchers want to learn more about these symptoms and find better ways to measure pain in people with NF1.

Objective:

To learn if a device called the AlgometRx Nociometer(Registered trademark) is effective in measuring pain or other abnormal sensations in people with NF1.

Eligibility:

People aged 1 year and older with NF1.

Design:

Individuals can have up to 3 assessments completed in person. Each assessment may last up to 1.0 to 1.5 hours.

Individuals will be screened. They will complete questionnaires about their health and how bad their pain is. If participants are having blood drawn for other reasons, some additional samples may be used in this study.

The AlgometRx Nociometer includes an electrode that will be placed onto a finger or a toe. The electrode will send non-painful electrical signals to activate nerves in the finger or toe. At the same time, a camera will be used to record changes in the pupil of the eye. The test will be done on all 4 of the participant s limbs; however, researchers may skip 1 or more limbs for various reasons. This test takes about 10 seconds to complete with at least a one-minute rest between testing different limbs.

Individuals will be asked to do a 2nd assessment with the AlgometRx Nociometer that may be done 1 hour later but no more than 72 hours after the first assessment. Participants who will be returning for another visit can opt to do a 3rd assessment that will be done at least 4 weeks but not more than 18 months after the 1st....

DETAILED DESCRIPTION:
Background:

* Chronic pain is a common and often debilitating symptom of neurofibromatosis 1 (NF1) that is related to multiple tumor (e.g., plexiform neurofibromas; PN) and non-tumor (e.g., headaches) manifestations.
* Patient-reported outcome (PRO) measures have been used to assess pain in PN trials; however, few are validated for NF populations. In addition, the subjective measurement of pain symptoms can be difficult particularly in young children, those with learning disabilities, and due to patients having various types of NF-related pain and other sensory problems.
* There is a critical unmet need for a simple, non-invasive, and objective measure of pain and other sensory problems for individuals with NF1.
* AlgometRx Nociometer (Registered Trademark) is a novel integration of infrared video pupillometry and neuroselective stimulation, and the outcome measure obtained from an assessment with this device is the Neuropathy Index. The use of the AlgometRx Nociometer (Registered Trademark) in studies was determined to be non-significant risk (NSR) by the Children s National Hospital (CNH) Institutional Review Board (IRB) based on similar technologies that have been defined by the Food and Drug Administration (FDA) to be NSR.
* In addition to the early detection and targeted clinical management and monitoring of pain and nociceptive processing in patients with NF1, this device also may help us learn more about the underlying mechanisms of their pain, as well as their symptoms of numbness and tingling (paresthesia), muscle weakness, loss of reflexes/hyperreflexia, and altered sensation.
* This novel biomarker could fill a critical gap for an objective, simple, and sensitive assessment to quantify and monitor NF-related pain as a physiologic measure for clinical monitoring and as potential surrogate marker for response in treatment trials.

Objective:

-To describe the feasibility of using the AlgometRx Nociometer (Registered Trademark) device to conduct a physiologic assessment of pain in different age groups of participants with NF1.

Eligibility:

* Participants must have a history of clinical or genetic diagnosis of NF1
* Age >= 1 year
* At least one eye with an intact pupillary reflex
* At least one digit (finger or toe) without open wounds for application of the device
* Must understand English or Spanish
* Participants who are < 18 years must have a caregiver willing to help the child engage in study procedures, assist with fitting the AlgometRx Nociometer (Registered Trademark) device, and complete the observer reported (ObsRO) measures. Note: the caregiver of a child participant >= 5 years old must be able to understand English or Spanish, the caregiver of a child participant 1-4 years old must be able to understand English (to help complete the observational pain measure for the younger children that is only available in English).

Design:

* The design will be a multi-site diagnostic pilot study to describe the feasibility and acceptability and to evaluate the initial psychometric properties (reliability, validity, sensitivity to change) of a novel objective pain measurement device [AlgometRx Nociometer (Registered Trademark)] for use in future clinical trials for participants with NF1. NCI is the lead site and Children's National Hospital (CNH) is the participating site; both sites will enroll participants with NF1 in this study.
* A cross-sectional design will be used to describe the acceptability of the assessment with the AlgometRx Nociometer (Registered Trademark) device as well as construct validity of the Neuropathy Index. A longitudinal design will be used to assess test-retest reliability and sensitivity to change of the Neuropathy Index.
* The sample will consist of 55 evaluable participants who will be placed into 5 cohorts defined by age (1-4; 5-7; 8-12; 13-17; >= 18 years) with approximately 11 participants in each group (plus/minus 3) and total enrollment of 70 participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* History of clinical or genetic diagnosis of NF1 as per the 2021 revised diagnostic criteria
* Age >= 1 year
* At least one digit (finger or toe) without open wounds for application of the device
* Individuals must understand English or Spanish
* Individuals who are < 18 years must have a caregiver willing to help the child engage in study procedures, assist with fitting the AlgometRx Nociometer (Registered Trademark) device, and complete the observer reported (ObsRO) measures. Note: the caregiver of a child participant >= 5 years old must be able to understand English or Spanish, the caregiver of a child participant 1-4 years old must be able to understand English (to help complete the observational pain measure for the younger children that is only available in English)
* Ability of individual or parent/guardian to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA

* History of eye pathology which precludes pupillometry, such as problems with pupillary reflex, blindness or inability to open at least one eye fully for evaluation
* Individuals with chronic use of medication that specifically affects their pupillary response, such as atropine-containing eye drops
* Uncontrolled intercurrent illness evaluated by medical history that would potentially increase in risk of participant

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Describe the feasibility of using AlgometRx Nociometer device in different age groups | Baseline (enrollment, Time 1)
  Proportion of individuals who successfully complete the AlgometRx Nociometer assessment by each of the five age stratified groups (1-4, 5-7, 8-12, 13-17, 18+ years). This analysis will be performed on the Feasibility Analysis Data Set. Successful completion rate for each age group.

SECONDARY OUTCOMES:
Describe the acceptability of the physiologic pain assessment using the AlgometRx Nociometer device in different age groups | Time 1
  Acceptability will be described per age group for the three questions on the Acceptability Questionnaire.
Evaluate the test-retest reliability of the physiologic pain measure (Neuropathy Index) | Time 1, repeated 1-72 hours later (Time 2)
  Test-retest reliability will be measured by the intraclass correlation coefficient in participants with stable pain.
Evaluate the construct validity of the physiologic pain measure (Neuropathy Index) | Time 1
  Convergent and discriminant validity with the PRO/ObsRO measures will be measured through parametric (Pearson s) or nonparametric (Spearman s) tests, depending on the normality and distribution of the data.
Evaluate the physiologic pain measure (Neuropathy Index) on sensitivity to change in pain | Time 1, repeated 4 weeks to 18 months later (Time 3)
  Sensitivity to change will be measured through paired t-tests or Wilcoxon signed-rank test, depending on the normality and distribution of the data, to evaluate the statistical significance of the change in scores. We also may use standardized response means, which is a type of effect size, and one of the best methods to estimate responsiveness of measures.
Evaluate safety of physiologic pain assessment | Time 1, Time 2, Time 3
  Evaluated by collection and assessment of ADEs (adverse device effects).

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Wolters, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001826-C.html